CLINICAL TRIAL: NCT01243996
Title: High-dose Ibuprofen for Patent Ductus Arteriosus in Extremely Preterm Infants: a Randomized Controlled Study
Brief Title: High-dose Ibuprofen for Patent Ductus Arteriosus (PDA) in Preterm Infant
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Carlo Dani, MD, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CD63-1
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-07

CONDITIONS: Ductus Arteriosus, Patent
Keywords: Patent ductus arteriosus, ibuprofen, preterm infants
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Infant treated with high dose ibuprofen (Experimental)
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — Treatment with high (20-10-10 mg/kg/day)or standard dose(10-5-5 mg/kg/day) ibuprofen
  Other Names: Pedea, Orphan Europe, Paris, France

SUMMARY:
The investigators hypothesized that the early treatment of PDA with ibuprofen doses higher than those actually recommended might increase the closure rate in preterm infants with gestational age <29 weeks without increasing the occurrence of associated adverse effects. To assess this hypothesis the investigators planned a multicenter randomized controlled study to compare the effectiveness of the current ibuprofen regimen to that of a high-dose regimen in closing PDA.

DETAILED DESCRIPTION:
The patency of ductus arteriosus (PDA) is a frequent complication in preterm infants suffering from respiratory distress syndrome (RDS), and 60% to 70% of preterm infants of <28 weeks' gestation receive medical or surgical therapy for a PDA [1]. Neonates with a left-to-right shunt through the ductus complicating their RDS have higher respiratory failure, lower survival rate, and increased risk of intracranial haemorrhage (ICH), bronchopulmonary dysplasia (BPD) and necrotizing enterocolitis (NEC) [2]. Therefore, closure of PDA is indicated before a significant left-to-right shunting occurs.

Patent ductus arteriosus can be treated effectively with intravenous indomethacin and ibuprofen, leading to permanent ductal closure in 60% to 80% of infants [3-5]. However, preterm infants treated with ibuprofen experience lower serum creatinine values, higher urine output, and less undesirable decreased organ blood flow and vasoconstrictive adverse effects than indomethacin-treated patients [4].

Recently, Sperandio et al. reported that high-doses of indomethacin (1 mg/kg: fivefold the usual dose) were safe and effective in closing PDA in 98.5% of infants with gestational age < 33 weeks, and demonstrated that the closure rate of PDA was related to the cumulative dose of given indomethacin [6]. Moreover, Desfrere et al. demonstrated that the currently recommended dose regimen of ibuprofen (10-5-5 mg/kg/day) is associated with a low estimated probability (30.6%) of closing PDA in infants while a high-dose regimen (20-10-10 mg/kg/day) might be associated with a greater, although unsatisfactory, probability (54.8%) of closing PDA, without relevant side affects [7]. Furthermore, Hirt et al., based on pharmacokinetic findings, proposed increasing the dose regimen of ibuprofen during the postnatal period from 10-5-5 mg/kg/day in preterm infants <70 h of age to 14-7-7 mg/kg/day in infants 70-108 h of age and 18-9-9 mg/kg/day in infants 108-180 h of age [8].

These studies [6-8] suggest that the failure of pharmacologic PDA closure might be due to the inadequacy of the standard dose regimen because of large interindividual pharmacokinetics and pharmacodynamic variations in premature infants during treatment for PDA [9,10].

The investigators hypothesized that the early treatment of PDA with ibuprofen doses higher than those actually recommended might increase the closure rate in preterm infants with gestational age <29 weeks without increasing the occurrence of associated adverse effects. To assess this hypothesis the investigators planned a multicenter randomized controlled study to compare the effectiveness of the current ibuprofen regimen to that of a high-dose regimen in closing PDA.

MATERIAL AND METHODS Patients Four tertiary neonatal intensive care units participated in the trial (the Careggi University Hospital of Florence, the Sant'Anna University Hospital of Turin, the Regional Hospital of Bozen, the IRCCS Ospedale Maggiore Policlinico of Milan). The study was approved by the medical ethics committee of each center. Neonates were enrolled after written informed consent was obtained from their parents.

The criteria for enrolment were a gestational age <29 weeks; an echocardiographic evidence of significant PDA; an age of 12 to 24 hours; and RDS necessitating respiratory support. Exclusion criteria were major congenital anomalies; life-threatening infection or hydrops fetalis; pulmonary hypertension; death before the conclusion of the first course of ibuprofen; urine output below 1 ml per kilogram of body weight per hour during the preceding 12 hours (with the exception of the first dose); a serum creatinine concentration of >1.5 mg/dL (129 μmol per liter); a platelet count of <50,000/mm3; a tendency to bleed, as revealed by hematuria, blood in the endotracheal aspirate, gastric aspirate, or stools, and oozing from puncture sites.

Study design The infants in each unit were randomly assigned to a treatment group by means of cards in sealed opaque envelopes. Each infant received three doses of intravenous ibuprofen (Pedea, Orphan Europe, Paris, France) either according to the standard regimen: an initial dose of 10 mg/kg, followed by two doses of 5 mg/kg each, after 24 and 48 hours; or at high-dose regimen: an initial dose of 20 mg/kg, followed by two doses of 10 mg/kg each, after 24 and 48 hours. The treatment was started at 12 to 24 hours of age and the medication was infused continuously over a period of 15 minutes.

When the ductus arteriosus was still patent after the randomly assigned treatment in a patient in either group a second course of ibuprofen at high-dose (20-10-10 mg/kg/day) was given as nonrandomized treatment, starting 24 hours after the last dose of the first course. If there was a contraindication to the second pharmacologic treatment, or if this therapy also failed to promote ductal closure, subsequent pharmacological and/or surgical treatment of PDA was at the discretion of the each center.

The plasma ibuprofen concentration was measured in blood samples obtained 15 minutes after the first dose of ibuprofen and 24 hours after the last dose 6 using high-pressure liquid chromatography (HPLC), as previously described [11].

Echocardiography The first heart ultrasound examination was performed at 12 to 24 hours of age to ascertain the normality of cardiac anatomy, to rule out the possibility of congenital heart disease with "ductus dependent" pulmonary or systemic blood flow and pulmonary hypertension, and to evaluate the PDA. The diagnosis of hemodynamically significant PDA requiring treatment was made by echocardiographic demonstration of a ductal left- to-right shunt, with a left atrium to aortic root ratio >1.3 or a ductal size >1.5 mm 12. In enrolled patients echocardiography was repeated after each dose of ibuprofen (12-24 hours after the last dose of the assigned treatment) and at 7+1, 15+2, 30+2 days of life to detect a possible re-opening of PDA. All echocardiographic studies were performed by physicians who were unaware of the infants' treatment assignments.

Fluid intake was guided by the body weight, serum sodium concentrations and serum osmolality. Daily fluid intake started with 70-80 ml per kilogram and was increased by 10-20 ml/kg/day up to 150 mL/kg at the end of the first week of life.

For treatment of RDS, infants received oxygen-therapy, respiratory supports (nasal continuous positive pressure, patient-triggered ventilation, high frequency oscillatory ventilation), and rescue surfactant treatment (Curosurf, Chiesi Farmaceutici Spa, Parma, Italy: first dose: 200 mg/kg; following dose: 100 mg/kg).

Gestational age, birth weight, sex, type of delivery, antenatal steroid treatment and main maternal pregnancy pathologies (preterm non-induced labor, hypertensive disorders, premature rupture of membranes, abruptio placentae, intrauterine growth restriction), highest FIO2 and mean airway pressure (MAP) values, type and duration of respiratory support, need of surfactant; daily fluid intake during the 1st week of life, and need of dopmine/dobutamine or plasma for hypotension were recorded for each infant. Serum creatinine was dosed at 1, 3, and 7 days of life, while daily urine output was measured through its collection in adhesive urine bags during the 1st week of life. Oliguria was defined as a urine output <1 ml/kg/h during a 24-hour collection period. Moreover, platelet count was measured at 1, 3, and 7 days of life and bleeding disorders (as revealed by hematuria, blood in the endotracheal aspirate, gastric aspirate, or stools, and oozing from puncture sites) were recorded during the 1st week of life.

For each infants were reported: the occurrence of ICH and ICH and periventricular hemorrhage (PVL) [13,14], BPD [15], retinopathy of prematurity (ROP) [16], NEC [17], sepsis [18], mortality and duration of hospitalization.

Statistical analysis The primary endpoint of the study was to evaluate the successful rate in closing PDA using ibuprofen. The investigators considered ibuprofen failure to be the lack of PDA closure at the end of the first course of ibuprofen in both the standard and high-dose regimen groups. On the basis of the data and in agreement with data from the literature 3-5, the investigators assumed a failure rate of 25% in the group treated with the standard ibuprofen regimen. Thus, to detect as statistically significant a decrease of failure rate of 20 % (to 5%) in the group treated with the high ibuprofen regimen, the investigators calculated that a sample size of at least 34 infants in each group was necessary at a power of 0.80 and α=0.05.

Clinical characteristics of the two groups were described by mean values and standard deviation, or median values and range, or by rate and percentage. The t-test, Wilcoxon rank-sum test, and Fisher's exact test were used to compare continuous normally distributed data, nonparametric continuous data, and categorical data, respectively.

Secondary endpoints were the evaluation of the effectiveness of the high-dose ibuprofen course in closing PDA refractory to the first ibuprofen course; possible association between dose regimen, occurrence of adverse effects, and ibuprofen plasma level; comparison of the incidence of ICH, PVL, ROP, NEC, BPD, sepsis, death and hospital stay duration in the two groups.

Multiple logistic regression was performed to assess the influence of predictive factors on the rate of PDA after the 1st ibuprofen course; the factors the investigators analyzed were gestational age, sex, birth weight, use or nonuse of antenatal glucocorticoid, highest FIO2 and MAP values, assignment to standard or high-dose ibuprofen regimen group. Effect estimates are expressed as relative risk (RR) with profile likelihood-based 95% confidence limits.

REFERENCES

1. Clyman RI. N Engl J Med 2000;343:728-30
2. Hamrick SE et al. Pediatrics 2010;125:1020-1030.
3. Itabashi K et al. J Pediatr 2003 ;143:203-207.
4. Thomas RL et al. Eur J Pediatr 2005;164:135-40.
5. Gournay V et al. Lancet. 2004;364:1939-44.
6. Sperandio M et al. Pediatrics 2005;116:1361-6.
7. Desfrere L etal. J Clin Pharm Ther 2005;30:121-32.
8. Hirt D et al. Br J Clin Pharmacol 2008;65:629-36.
9. Van Overmeire B et al. Clin Pharmacol Ther 2001;70:336-43.
10. Seybert HP et al. Eur J Pediatr 1983;141:71-6.
11. Rey E et al. British Journal of Clinical Pharmacology 1994;38:373-5.
12. Varvarigou A et al. JAMA 1996;275:539-44.
13. Papile LS et al. J Pediatr 1978;92 :529-34.
14. De Vries LS et al. Beha Brain Res 1992;49:1-6.
15. Ehrenkranz RA et al. Pediatrics 2005;116:1353-60.
16. Committee for the Classification of the Retinopathy of Prematurity. Arch Ophthalmol 1984;102:1130-4.
17. Bell MJ et al.Ann Surg 1978;187:1-12.
18. American Academy of Pediatric's Committee on drugs, Committee on fetus and newborn and Committee on Infectious Diseases. Pediatrics 1980;65:1047-53.

ELIGIBILITY:
Inclusion Criteria: Gestational age <29 weeks; an echocardiographic evidence of significant PDA; an age of 12 to 24 hours; and RDS necessitating respiratory support.

-

Exclusion Criteria: Major congenital anomalies; life-threatening infection or hydrops fetalis; pulmonary hypertension; death before the conclusion of the first course of ibuprofen; urine output below 1 ml per kilogram of body weight per hour during the preceding 12 hours (with the exception of the first dose); a serum creatinine concentration of >1.5 mg/dL (129 μmol per liter); a platelet count of <50,000/mm3; a tendency to bleed, as revealed by hematuria, blood in the endotracheal aspirate, gastric aspirate, or stools, and oozing from puncture sites.

-

Ages: 12 Hours to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2008-06; Primary Completion 2010-05 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Successful rate in closing PDA of ibuprofen administered at high or standard dose. | Between 84 and 96 hours of life

SECONDARY OUTCOMES:
Effectiveness of a second high dose ibuprofen course; correlation between peak plasma level of ibuprofen and PDA closure; mortality or BPD among survivors, incidence of ICH, PVL, ROP, NEC, sepsis, and length of stay in hospital. | Hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Dani, MD, Study Chair — University of Florence, Italy
Locations (1):
- Careggi University Hospital, Division of Neonatology, Florence, Italy

REFERENCES:
- [Derived] Dani C, Vangi V, Bertini G, Pratesi S, Lori I, Favelli F, Ciuti R, Bandinelli A, Martano C, Murru P, Messner H, Schena F, Mosca F. High-dose ibuprofen for patent ductus arteriosus in extremely preterm infants: a randomized controlled study. Clin Pharmacol Ther. 2012 Apr;91(4):590-6. doi: 10.1038/clpt.2011.284. Epub 2011 Nov 16. PMID 22089267